CLINICAL TRIAL: NCT03164252
Title: Low Power Laser in the Second Molar Tissue Repair and in the Postoperative of Mandibular Third Molar Surgery - Double Blind Randomized Clinical Trial.
Brief Title: Low Power Laser in Mandibular Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Michelle Bianchi de Moraes, Professor Assistente Doutor - Departamento de Diagnóstico e Cirurgia - São Paulo State University (Unesp), Institute of Science and Technology, São José dos Campos, Brasil., Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 47325515.3.0000.0077
Record Dates: First submitted 2017-05-18; First posted 2017-05-23 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Laser Therapy, Low-Level
Keywords: Third molar;; Third molar surgery;; Laser;; Tissue Repair.
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The sample of this study will be composed of 60 patients between 16 and 40 years old, who need to undergo the extraction of third molars included and / or impacted. The patients will be those who voluntarily seek the Discipline of Buccomaxillofacial Surgery and Traumatology, at the State University of São Paulo "Júlio de Mesquita Filho" - Unesp, to perform the procedure.
  This study will be a randomized, double-blind, prospective clinical trial with the following groups:
  Group I (with 20 patients) - laser therapy used in the immediate postoperative period will be intraoral irradiation with 660 nm red diode laser, 30 mW power and 10 J / cm2 fluency.
  Group II (with 20 patients) - laser therapy used in the immediate postoperative period will be intraoral irradiation with 660 nm red diode laser, 30 mW power and 30 J / cm2 fluency.
  Group III (with 20 patients) - Control Group - Application of laser sham.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Surgical procedures were always performed by the same surgeon and assistant, who were unaware of the surrogate group that belonged to the patient, as well as the patient himself. This randomization was performed involving numbers and envelopes, being only the investigator's knowledge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Grupo I- Lower laser fluency (Active Comparator): 20 patients received 660 nm red laser diode laser therapy, 30 mW power and 10 J / cm2 fluency, in the immediate period after surgical period of the third molar third molar extraction / impacted by the intraoral region
  Interventions: Radiation: Grupo II- Greater laser fluency; Radiation: Grupo III- Laser sham
- Grupo II- Greater laser fluency (Active Comparator): 20 patients received 660 nm red laser diode laser therapy, 30 mW power and 30J / cm2 fluency, in the immediate period after surgical of the third molar third molar extraction / impacted by the intraoral region
  Interventions: Radiation: Grupo I- Lower laser fluency; Radiation: Grupo III- Laser sham
- Grupo III- Laser sham (Placebo Comparator): Application of laser sham, the handpiece of the device will be positioned intraorally and activated. However, the tip of the applicator will be covered by an opaque material that prevents radiation from passing through.
  Interventions: Radiation: Grupo I- Lower laser fluency; Radiation: Grupo II- Greater laser fluency

INTERVENTIONS:
Radiation: Grupo I- Lower laser fluency — The region determined for the application of the laser will be 4 points of the gingival mucosa: 1 - center of the alveolus; 2- center of the cervical third of the lingual face; 3 - lingual face; And 4 - apical third of the lingual face. The application time of the laser will be divided equally between the four points of application.
  Other Names: Red laser diode of 660 nm/ power 30 mW/ creep of 10 J / cm2
  Arms: Grupo II- Greater laser fluency; Grupo III- Laser sham
Radiation: Grupo II- Greater laser fluency — The region determined for the application of the laser will be 4 points of the gingival mucosa: 1 - center of the alveolus; 2- center of the cervical third of the lingual face; 3 - lingual face; And 4 - apical third of the lingual face. The application time of the laser will be divided equally between the four points of application.
  Other Names: Red laser diode of 660 nm/ power 30 mW/ creep of 30 J / cm2.
  Arms: Grupo I- Lower laser fluency; Grupo III- Laser sham
Radiation: Grupo III- Laser sham — The region determined for the application of the laser will be 4 points of the gingival mucosa: 1 - center of the alveolus; 2- center of the cervical third of the lingual face; 3 - lingual face; And 4 - apical third of the lingual face. The application time of the laser will be divided equally between the four points of application.
  Other Names: Control group, application of laser sham
  Arms: Grupo I- Lower laser fluency; Grupo II- Greater laser fluency

SUMMARY:
The low-power laser provides the body with an improvement in the inflammatory response. Thus, the objective of this study is to evaluate two laser application protocols in 60 patients requiring surgical treatment for extraction of third molars included, without distinction of race or gender, aged between 16 and 40 years, coming from the Faculty of Dentistry Of São José dos Campos (UNESP). These patients will be divided randomly into 3 groups: group 1 - intraoral irradiation with 660 nm laser at a dose of 10 J (30 mW, 10 J / cm 2) , group 2 - intraoral irradiation with 660 nm laser at a dose of 30 J (30 mW, 30 J / cm 2) and group 3- control group, with application of placebo laser. At 3 and 7 days after surgery, the patients will be evaluated by two evaluators who will measure edema, trismus and pain. The tissue repair will also be evaluated after 1, 3 and 6 months of surgery, through radiographic analysis and periodontal conditions in the distal of the lower second molar. The results will be submitted to descriptive statistics and compared using the statistical analysis of variance (ANOVA) and Tukey test with significance level of 5%.

DETAILED DESCRIPTION:
Knowing the ability of the low-power laser to provide the body with an improvement in inflammatory response, with consequent reduction of edema, minimizing painful symptoms and leading to biostimulation, laser therapy is presented as an alternative for processes that present an inflammatory reaction, Pain and need for tissue regeneration. The literature shows the efficacy of laser in the postoperative surgery for extraction of third molars. However, to date, there is no consensus on the best protocol to be used in these cases. Thus, the objective of this study will be to evaluate two laser application protocols. To this end, 60 patients will be selected who require surgical treatment for the extraction of third molars, regardless of race or gender, between the ages of 16 and 40, from the School of Dentistry of São José dos Campos (UNESP). These patients will be divided randomly into 3 groups: group 1 - intraoral irradiation with 660 nm laser at a dose of 10 J (30 mW, 10 J / cm 2), group 2 - intraoral irradiation with 660 nm laser at a dose of 10 J (30 mW, 10 J / cm 2) and group 3 - control group, with application of placebo laser. At 3 and 7 days after surgery, patients will be evaluated by two evaluators who will measure edema, mouth opening (assessment of muscle spasm) and pain. To compare the data, we will use the analog pain scale (VAS), the method of Ustün et al. (2003), and the millimeter rule. The patient will also be questioned about possible postoperative problems, as well as the surgeon, who will classify the postoperative repair process according to Batinjan et al. (2013). The tissue repair will also be evaluated after 1, 3 and 6 months of surgery, through radiographic analysis and periodontal conditions in the distal of the lower second molar. The results will be submitted to descriptive statistics and compared using the statistical analysis of variance (ANOVA) and Tukey test with significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients, without surgical contraindications, requiring avulsion of the included third molars and / or impacted lower molars,
* Teeth classified according to Winter (1926) as mesioangulated and according to Pell & Gregory (1933) as 1A to 2B.
* Between the ages of 16 and 40
* Who have agreed to participate in the research voluntarily, after knowing the risks and benefits, and signed the Informed Consent Term (TCLE)

Exclusion Criteria:

* Patients with any systemic or local change that contraindicate the procedure,
* Use of anti-inflammatories in the last 15 days,
* Patients smokers or diabetics.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2016-12-06 (Actual)

PRIMARY OUTCOMES:
Periodontal probing | Initially carried out in one, three and six months
  Evaluated in patients in groups I (Lower laser fluency), II (Greater laser fluency) and III (Laser sham). For the investigator periodontal evaluation was performed based on the modified Montero & Mazzaglia (2011) methodology, where the length of the clinical crown in the second distal molar region will be measured with a North Carolina-type probe (Hu-Friedy, Chicago, USA). According to this methodology, we will previously mold the occlusal of the second molar with a condensation silicone (Optosil Xantopren, Heraeus Kulzer, Hanau, Germany), which was used as a guide to standardize the location and height of the measurement. We will then measure at three points in the distal of the second molar: disto-lingual, mesio-distal and vestibular-distal.

SECONDARY OUTCOMES:
Pain assessment | Evaluated immediately, two, four, six and eight hours after surgery. And with continuity for one, two, three and four days
  Evaluated in patients in groups I (Lower laser fluency), II (Greater laser fluency) and III (Laser sham).The investigators were based on the analogue pain scale (VAS).
Edema assessment | Initially carried out in three and seven days.
  Evaluated in patients in groups I (Lower laser fluency), II (Greater laser fluency) and III (Laser sham). For investigators to measure facial edema used the method of Ustün et al. (2003) and a millimeter rule to obtain the measures.
Trismus assessment | Initially carried out in three and seven days
  Evaluated in patients in groups I (Lower laser fluency), II (Greater laser fluency) and III (Laser sham). To measure the buccal opening, the distance between the incisal edges of the maxillary and mandibular incisors, obtained with the patient sitting upright, will be evaluated by a millimeter ruler.
Radiographic assessment | Assessment in one, three and six months
  Evaluated in patients in groups I (Lower laser fluency), II (Greater laser fluency) and III (Laser sham). Radiographic evaluation will be performed using the methodology as recommended by Ogundipe et al. (2011), who performed periapical radiographs of the investigators region and classified the bone repair based on three variables: hard blade, bone density and trabecular pattern according to a specific table.

OTHER OUTCOMES:
Tissue repair | Assessment in three days
  Evaluated in patients in groups I (Lower laser fluency), II (Greater laser fluency) and III (Laser sham).The surgeon through the methodology proposed by Batinjan et al. (2013), will classify four indirect variables.
Problems encountered after surgery | Assessment in four days
  Evaluated in patients in groups I (Lower laser fluency), II (Greater laser fluency) and III (Laser sham). The patients evaluated indirectly through the methodology proposed by Batinjan et al. (2013) with the completion of three variables.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle B Moraes, PHD, Principal Investigator — ICT-Unesp

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lago-Mendez L, Diniz-Freitas M, Senra-Rivera C, Gude-Sampedro F, Gandara Rey JM, Garcia-Garcia A. Relationships between surgical difficulty and postoperative pain in lower third molar extractions. J Oral Maxillofac Surg. 2007 May;65(5):979-83. doi: 10.1016/j.joms.2006.06.281. PMID 17448851
- [Result] Lopez-Ramirez M, Vilchez-Perez MA, Gargallo-Albiol J, Arnabat-Dominguez J, Gay-Escoda C. Efficacy of low-level laser therapy in the management of pain, facial swelling, and postoperative trismus after a lower third molar extraction. A preliminary study. Lasers Med Sci. 2012 May;27(3):559-66. doi: 10.1007/s10103-011-0936-8. Epub 2011 May 27. PMID 21617973
- [Result] Montero J, Mazzaglia G. Effect of removing an impacted mandibular third molar on the periodontal status of the mandibular second molar. J Oral Maxillofac Surg. 2011 Nov;69(11):2691-7. doi: 10.1016/j.joms.2011.06.205. Epub 2011 Aug 23. PMID 21864969